CLINICAL TRIAL: NCT02306005
Title: Insulin Therapy and Quantitive and Qualitive Changes of Plasma Lipoproteins in Patients With Newly Diagnosed Type 1 Diabetes.
Brief Title: Insulin Therapy and Lipoproteins' Profile in Type 1 Diabetes.
Acronym: InLipoDiab1
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aleksandra Uruska, PhD, MD, Poznan University of Medical Sciences
Other Study IDs: 856/14
Record Dates: First submitted 2014-11-23; First posted 2014-12-03 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes mellitus type 1, insulin therapy, lipoproteins, HDL
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 diabetic patients: Newly diagnosed diabetes type 1 admitted to the Department of Internal Medicine and Diabetology. Measurement of lipid profile and lipoproteins before and after administration of insulin. Further continuous observation with follow-up every year and evaluation of final end-points after 5 and 10 years.

SUMMARY:
The aim of the study is to evaluate the effect of insulin therapy in patients with newly diagnosed type 1 diabetes on quantitative and qualitative changes of plasma lipoproteins, with particular emphasis on HDL metabolism, and analysis of the factors determining the effect of insulin therapy on lipid profile.The study is planned to cover a minimum of 100 people with newly diagnosed type 1 diabetes and lead prospective observation of this group (for a minimum of 5-10 years). Patients will be assessed: during the first hospitalization in the moment of diagnosis (prior to introduction of insulin treatment), after 3 weeks, after 6 months and after 12 months of insulin therapy. Further observations planned in the annual intervals. In addition, the study group will be under constant monitoring of metabolic evaluation every three months in the Outpatient Clinic.

During each follow-up will be assessed parameters evaluating the metabolism of plasma lipoprotein fractions and subfractions of HDL:

1. The concentration of apolipoprotein: including A-I, A-II, A-IV, C (II and III), D and E
2. Electrophoresis of plasma lipoproteins
3. Electrophoresis of HDL
4. The activity of enzymes: acyltransferase lecithin: cholesterol (LCAT) and plasma lipoprotein lipase Moreover, evaluation of factors which may potentially modify the relation between insulin therapy and lipoproteins will be assessed

   1. Anthropometric data and markers of insulin resistance (such as BMI, waist-hip ratio, the estimated rate of glucose distribution, VAI index, body fat, blood pressure),
   2. Metabolic management of diabetes,,
   3. Protein glycation end products
   4. The concentration of plasma adipokines.

Expected impact of the research project on the development of science, civilization and society The obtained results allow to assess the impact of exogenous insulin on quantitative and qualitative changes and metabolism of lipoproteins in the serum of patients with type 1 diabetes. Understanding the etiopathogenesis of this phenomenon and the factors affecting it seem to be very important in the treatment of patients with type 1 diabetes, where insulin is the treatment of choice and dosage adjustment appears to be extremely important. Remains unknown whether the changes in the lipoprotein profile result from the beginning of insulin therapy or other factors influence it. Selecting a group of patients with less favorable lipoprotein profile may allow better metabolic control, and thus will affect the quality and length of life of our patients. These studies will assess the impact of our therapeutic actions on the diagnosis of the disease on long-term consequences, such as the development of chronic complications.

ELIGIBILITY:
Inclusion Criteria:

* New onset type 1 diabetes and treatment with insulin.
* Written consent to participate in the study.
* There are no other medical conditions, and with no other additional drugs beyond insulin

Exclusion Criteria:

* any other medical conditions, and any other additional drugs beyond insulin

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A minimum of 100 people with newly diagnosed type 1 diabetes hospitalized in the Department of Internal Medicine and Diabetology Poznan University of Medical Sciences
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Changes in lipoproteins' metabolism | Change from Baseline in lipoproteins' metabolism at 6 and 12 months
  Evaluation of HDL levels, subfractions and enzymes connected with HDL metabolism (LCAT, lipoprotein lipase)
Factors influencing relationship between insulin treatment and lipoproteins | 1 year
  Metabolic control, presence of remission, insulin resistance, adipokines, daily insulin requirement

SECONDARY OUTCOMES:
Changes in apolipoproteins | Change from baseline in apolipoproteins' at 6 and 12 months
  Evaluation of apolipoproteins: A-I, A-II, A-IV, C (II i III), D i E
Presence of insulin resistance | 1 year
  Evaluation of lipid tissue content, VAI, triglycerides/HDL ratio and estimated glucose disposal rate
Development of Retinopathy | 1 year
  Evaluation of retinopathy (ophthalmology assessment)
Development of Neuropathy | 1 year
  Evaluation of presence of neuropathy peripheral and autonomic (clinical examination and ProsciCard)
Development of Diabetic kidney disease | 1 year
  Evaluation of presence of diabetic kidney disease (albuminuria, GFR)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine and Diabetiology Poznan University of Medical Sciences, Poznan, Poland

REFERENCES:
- [Result] Cieluch A, Uruska A, Grzelka-Wozniak A, Niedzwiecki P, Flotynska J, Zozulinska-Ziolkiewicz D. Changes in high-density lipoprotein cholesterol (HDL-C) level and the ratio of triglycerides to HDL-C during the first year of type 1 diabetes. Pol Arch Intern Med. 2019 Sep 30;129(9):598-604. doi: 10.20452/pamw.14920. Epub 2019 Aug 5. PMID 31379357
- [Result] Cieluch A, Uruska A, Grzelka A, Zozulinska-Ziolkiewicz D. An increase in high-density lipoprotein cholesterol concentration after initiation of insulin treatment is dose-dependent in newly diagnosed type 1 diabetes. The results of the InLipoDiab1 study. Pol Arch Intern Med. 2018 Jan 31;128(1):69-71. doi: 10.20452/pamw.4183. Epub 2018 Jan 19. No abstract available. PMID 29350676
- [Derived] Uruska A, Mietkiewska-Dolecka M, Grzelka-Wozniak A, Flotynska J, Saldanha S, Rohatgi A, Zozulinska-Ziolkiewicz D. Clinical remission in newly diagnosed type 1 diabetes mellitus and HDL function on cholesterol efflux capacity: prospective InLipoDiab1 study. Endocr Connect. 2025 Jun 17;14(6):e240704. doi: 10.1530/EC-24-0704. Print 2025 Jun 1. PMID 40465557